CLINICAL TRIAL: NCT04186455
Title: Comparison of Pro Seal and Baska-mask
Brief Title: Comparison of Laryngeal Masks in Urethral Cystoscopic Surgery Operations: a Prospective Randomized Clinical Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, Zehra Ipek ARSLAN, Associate Professor, Kocaeli University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: KAEK 2019/68
Record Dates: First submitted 2019-11-28; First posted 2019-12-04 (Actual); Last update posted 2022-02-08 (Actual); Status verified 2022-02

CONDITIONS: Ureteral Calculi
Keywords: baska-mask; proseal; urs
MeSH Terms: conditions — Ureteral Calculi | interventions — Laryngeal Masks

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- insertion time (Active Comparator): lma pro seal and basks-mask in patients undergoing ups
  Interventions: Device: proseal; Device: baska-mask
- oropharyngeal leak pressure (Active Comparator): lma baska-mask undergoing urs
  Interventions: Device: proseal; Device: baska-mask

INTERVENTIONS:
Device: proseal — laryngeal mask proseal
  Other Names: laryngeal mask
Device: baska-mask — laryngeal mask baska-mask
  Other Names: laryngeal mask

SUMMARY:
The use of Laryngeal masks are increased.This study aimed to compare lma pro seal and baska -mask in urethral retrograde sistoscopy operations.

DETAILED DESCRIPTION:
The use of Laryngeal masks are increased. Aimed to compare lma pro seal and baska -mask in urologic retrograde sistoscopy operations. ASA 1-2 80 subjects who is undergoing elective URS operations were enrolled in this prospective randomized clinical study. The demographic and airway characteristics of patients preoperatively and lam insertion times, nasogastric insertion times number of intubation attempts, fiberoptic grades from the lam, expired tidal volume, oropharyngeal leak pressures, peak and mean airway pressures preoperatively, minor complications like sore throat, hoarseness, dysphagia were recorded at the postoperative care unit.

ELIGIBILITY:
Inclusion Criteria:18-65 years of age

* undergoing elective urs operations
* bmı<35
* ASA I-II

Exclusion Criteria:<18 years of age

* bmı>35
* ASA III-IV

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2019-12-05 (Actual); Primary Completion 2022-02-07 (Actual); Study Completion 2022-02-07 (Actual)

PRIMARY OUTCOMES:
insertion time | 20 seconds
  insertion time of the laryngeal mask

CONTACTS AND LOCATIONS:
Locations (1):
- Kocaeli University Medical Faculty, Kocaeli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No